CLINICAL TRIAL: NCT00393341
Title: Quantitation of Endothelial Progenitor Cells as Markers of Tumor Angiogenesis in Breast Cancer
Acronym: EPC
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Kathy Miller, Ballve Lantero Professor of Oncology, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 0609-21; IUCRO-0168
Record Dates: First submitted 2006-10-25; First posted 2006-10-27 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer Stage IV; Breast Cancer Stage I; Breast Cancer Stage II
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample

GROUPS / COHORTS (2):
- Case: Women with breast cancer
  Interventions: Procedure: Blood Draw
- Control: Women without breast cancer
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Blood sample will be drawn from a vein in the arm.

SUMMARY:
We propose to quantitate endothelial progenitor cells (EPCs) in early and advanced breast cancer patients. Peripheral blood will be drawn from the eligible patients. Different type of EPCs will be isolated from the blood and quantitated.

DETAILED DESCRIPTION:
Accumulating evidence emphasizes the emerging role of circulating endothelial cells (CECs) and endothelial progenitor cells (EPCs) in tumor angiogenesis as surrogate markers and in the efficacy of anti-angiogenic therapies in breast cancer (22-27). Furstenberger et al. (22) reported that CECs were significantly elevated in breast cancer patients and decreased during chemotherapy (anthracycline and/or taxane based). However, EPCs (CD34+/VEGFR-2+) as well as their progenitor cell population CD133+/CD34+ and the population of CD34+ stem cells increased together with VEGF, erythropoietin and angiopoietin-2 levels. Their data suggest that chemotherapy reduces mature CECs, while mobilizing the EPC population. Using real-time PCR and flow cytometry, they also showed that CD146, an endothelial cell specific antigen, was significantly increased in newly diagnosed breast cancer patients compared to healthy controls (23). Other studies also reported increased circulating EPCs in breast cancer patients in addition to CECs (24,25). In another study, circulating EPCs were not increased in cancer patients despite the high plasma VEGF levels (26). Another interesting aspect is that Mancuso et al (27) showed that CEC kinetics correlate with progression-free and overall survival but not circulating progenitor cells in metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic breast cancer(stage IV), or women with a history of Stage I or II breast cancer disease who are currently disease free Women greater than or equal to 18 years of age Ability to understand and the willingness to sign an informed consent

Exclusion Criteria:

* Chemotherapy, radiation, or surgery within the past 4 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 18 or older with breast cancer recieving treatment at IUSCC and willing to donate a blood sample and complete consent form.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2006-10; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To quantitate endothelial progenitor cells (EPCs) in early and advanced breast cancer patients. Different type of EPCs will be isolated from the blood and quantitated. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: George W Sledge, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States